CLINICAL TRIAL: NCT01822665
Title: A Study to Investigate the Gastrointestinal Safety of OTC Analgesics in Healthy Volunteers by Endoscopic Examination
Brief Title: Gastrointestinal Safety Evaluation of Two Over the Counter Analgesics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A1901106
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2013-07

CONDITIONS: Gastrointestinal Mucosal Damage
MeSH Terms: interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Paracetamol Tablet (Active Comparator): Paracetamol 500 mg tablet, 2 tablets administered 4 times a day (QID) with water.
  Interventions: Drug: Paracetamol
- Ibuprofen Tablet (Active Comparator): Ibuprofen 400 mg tablet, 2 tablets administered three times a day (TID) with water
  Interventions: Drug: Ibuprofen
- Placebo Tablet (Placebo Comparator): Placebo tablets, 2 tablets QID administered with water.
  Interventions: Other: Placebo
- Ibuprofen Capsule (Active Comparator): Ibuprofen 400 mg liquid gel capsules, 2 tablets, TID administered with water
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Liquid gelation capsules or tablets of 400 mg strength
  Arms: Ibuprofen Capsule; Ibuprofen Tablet
Drug: Paracetamol — Paracetamol fast dissolving tablets of 500 mg strength
  Arms: Paracetamol Tablet
Other: Placebo — Placebo tablets
  Arms: Placebo Tablet

SUMMARY:
This study evaluated the effect of oral fast-dissolving formulations of paracetamol and ibuprofen on the lining of the stomach and duodenum (gastrointestinal mucosa). Endoscopic examinations were conducted to determine the gastrointestinal damage produced post a 7 day treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: 18-30 kg/m^2
* Body Weight 60-80 kg
* Participant with both a normal stomach and proximal duodenum mucosa as evidenced by endoscopic results

Exclusion Criteria:

* Participant with evidence of current/active, or a history of gastrointestinal disease
* Participant with a history of renal disease, pulmonary edema, cardiomyopathy, liver disease, intrinsic coagulation defects, bleeding diseases or anticoagulant therapy
* Participant with a history of using antacids, H2 receptor antagonists, proton pump inhibitors, or misoprostol more than twice a month or has used any of these medications within 1 week of Visit 1.
* Participant with a current or recurrent disease, within 12 months of Visit 1, that could affect the action, absorption, disposition, or excretion of the study treatments or evaluation of the clinical or laboratory tests

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Houston Institute for Clinical Research, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Of 41 participants screened, 12 did not meet the study criterion and one participant withdrew consent. Remaining 28 participants were randomized into the study to received all the four treatments in a sequential manner.
Groups:
- Overall Study: This was a randomized, 4-way crossover study. Participants received two fast dissolving paracetamol tablets (500 milligrams [mg]/tablet) four times daily (QID); two liquid-filled gelatin capsules containing ibuprofen (200 mg/capsule), three times daily (TID); two ibuprofen tablets (200 mg/tablet), TID; and, two fast dissolving placebo tablets QID. All the treatments were administered orally with water. There was a washout period of 7 days following every treatment session.
Period: Overall Study
Arm/Group | Overall Study
Started | 28
Received Ibuprofen Tablet (400 mg) | 23 (5 participants did not complete; Period 3(2:adverse events;1:other reason); Period 4(2:other reason))
Received Placebo Tablet | 23 (5 participants did not complete; Period 2(1:other reason); Period 4(3:adverse event; 1:other reason))
Received Ibuprofen Capsule (400 mg) | 24 (Two participants, each in period 3 and period 4 did not complete treatment for 'other reason'.)
Received Paracetamol Tablet (1000 mg) | 28
Completed | 20
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — Other Reason | 5

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants in the study who took at least one treatment dose.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.1 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Gastromucosal Damage (GMD) Score of Paracetamol Tablet vs Ibuprofen Capsule
Description: Endoscopic examination of the upper gastrointestinal mucosa evaluated the extent of mucosal injury to the stomach and the duodenum separately using a 5-point Lanza scale, ranging from 0: normal stomach; 1: mucosal hemorrhages; 2: one or two erosions; 3: numerous areas of erosions; and 4: more than 10 erosions or ulcer.
Time Frame: Day 7
Population: Intent to Treat (ITT) population: all participants who fulfilled all the study entry criteria and receive at least one of the study treatments. The ITT population included all participants with valid data-period. Missing data was not imputed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Paracetamol Tablet (1000 mg): Two paracetamol tablets (500 mg/tablet) was administered QID, orally with water.
- Ibuprofen Capsule (400 mg): Two ibuprofen capsules (400 mg/tablet), was administered TID, orally with water.
Arm/Group | Paracetamol Tablet (1000 mg) | Ibuprofen Capsule (400 mg)
Number analyzed (Participants) | 27 | 23
Scores on a scale | 0.33 (0.68) | 1.48 (1.34)
Statistical Analysis 1: Comparison: Paracetamol Tablet (1000 mg) vs Ibuprofen Capsule (400 mg); Null hypothesis considered no significant difference in mean endoscopy score of gastric mucosal damage between two treatments; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — No multiple comparisons were carried out; Period and treatment were included in the model as fixed effects, while subjects were a random effect; Least squares mean difference = -1.11, 95% CI 2-sided [-1.63 to -0.59] — Difference was first named treatment minus second named treatment, such that a positive difference favors the first named treatment

2. Secondary Outcome: GMD Scores of Paracetamol Tablet; Ibuprofen Capsule; Ibuprofen Tablet; and Placebo Tablet
Description: as for outcome 1
Time Frame: Day 7
Population: ITT population: All participants who fulfilled all the study entry criteria and received at least one of the study treatments. The ITT population included all participants with valid data-period. Missing data was not imputed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Paracetamol Tablet (1000 mg): Two paracetamol tablets (500 mg/tablet) were administered QID, orally with water.
- Ibuprofen Capsule (400 mg); Ibuprofen Tablet (400 mg): Two ibuprofen capsules (400 mg/tablet), were administered TID, orally with water.
- Placebo Tablet: Two placebo tablets were administered QID, orally with water.
Arm/Group | Paracetamol Tablet (1000 mg) | Ibuprofen Capsule (400 mg) | Ibuprofen Tablet (400 mg) | Placebo Tablet
Number analyzed (Participants) | 27 | 23 | 22 | 23
Score on a scale | 0.33 (0.68) | 1.48 (1.34) | 1.05 (1.33) | 0.14 (0.35)
Statistical Analysis 1: Comparison: Paracetamol Tablet (1000 mg) vs Ibuprofen Tablet (400 mg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0095, t-test, 2 sided; Period and treatment were included in the model as fixed effects, while subjects were a random effect; LS Mean Difference = -0.70, 95% CI 2-sided [-1.23 to -0.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Paracetamol Tablet (1000 mg) vs Placebo Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4794, t-test, 2 sided — No multiple comparisons were carried out; Period and treatment were included in the model as fixed effects, while subjects were a random effect; LS mean difference = 0.19, 95% CI 2-sided [-0.34 to 0.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Ibuprofen Capsule (400 mg) vs Ibuprofen Tablet (400 mg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1429, t-test, 2 sided — No multiple comparisons were carried out; Period and treatment were included in the model as fixed effects, while subjects were a random effect; LS mean difference = 0.40, 95% CI 2-sided [-0.14 to 0.95] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Ibuprofen Capsule (400 mg) vs Placebo Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — No multiple comparisons were carried out; Period and treatment were included in the model as fixed effects, while subjects were a random effect; LS mean difference = 1.30, 95% CI 2-sided [0.75 to 1.84] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Ibuprofen Tablet (400 mg) vs Placebo Tablet; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0020, t-test, 2 sided — No multiple comparisons were carried out; Period and treatment were included in the model as fixed effects, while subjects were a random effect; LS mean difference = 0.89, 95% CI 2-sided [0.34 to 1.45] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Duodenal Mucosal Damage (DMD) Scores
Description: DMD was measured using a 5- point Lanza scale: 0 - normal duodenum; 1 - mucosal hemorrhages; 2 - one or two erosions; 3 - numerous areas of erosions and 4 - more than 10 erosions/ ulcers.
Time Frame: Day 7
Population: ITT population: All participants who fulfilled all the study entry criteria and receive at least one of the study treatments. The ITT population included all participants with valid data-period. Missing data was not imputed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Ibuprofen Tablet (400 mg): Two ibuprofen tablets (400 mg/tablet), were administered TID, orally with water.
Arm/Group | Paracetamol Tablet (1000 mg) | Ibuprofen Capsule (400 mg) | Ibuprofen Tablet (400 mg) | Placebo Tablet
Number analyzed (Participants) | 27 | 23 | 22 | 23
Score on a scale | 0.15 (0.77) | 0.26 (0.86) | 0.23 (0.75) | 0.00 (0.00)
Statistical Analysis 1: Comparison: Paracetamol Tablet (1000 mg) vs Ibuprofen Capsule (400 mg); Null hypothesis considered no significant difference in mean endoscopy score of duodenal mucosal damage between two treatments; Test type: Superiority or Other; p = 0.6497, t-test, 2 sided — No multiple comparisons were carried out; Period and treatment were included in the model as fixed effects, while subjects were a random effect; LS mean difference = -0.09, 95% CI 2-sided [-0.49 to 0.31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Paracetamol Tablet (1000 mg) vs Ibuprofen Tablet (400 mg); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.7591, t-test, 2 sided — No multiple comparisons were carried out; Period and treatment were included in the model as fixed effects, while subjects were a random effect; LS mean difference = -0.06, 95% CI 2-sided [-0.46 to 0.34] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Paracetamol Tablet (1000 mg) vs Placebo Tablet; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.4126, t-test, 2 sided — No multiple comparisons were carried out; Period and treatment were included in the model as fixed effects, while subjects were a random effect; LS mean difference = 0.17, 95% CI 2-sided [-0.24 to 0.57] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Ibuprofen Capsule (400 mg) vs Ibuprofen Tablet (400 mg); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8903, t-test, 2 sided — No multiple comparisons were carried out; Period and treatment were included in the model as fixed effects, while subjects were a random effect; LS mean difference = 0.03, 95% CI 2-sided [-0.39 to 0.45] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Ibuprofen Capsule (400 mg) vs Placebo Tablet; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2227, t-test, 2 sided — No multiple comparisons were carried out; Period and treatment were included in the model as fixed effects, while subjects were a random effect; LS mean difference = 0.26, 95% CI 2-sided [-0.16 to 0.67] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Ibuprofen Tablet (400 mg) vs Placebo Tablet; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2855, t-test, 2 sided — No multiple comparisons were carried out; Period and treatment were included in the model as fixed effects, while subjects were a random effect; LS mean difference = 0.23, 95% CI 2-sided [-0.20 to 0.65] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Incidence of Gastric and/or Duodenal Mucosal Injury
Description: Number of participants with endoscopy score equal to or more than 2 were determined based on Lanza score for both gastric and duodenal mucosal damage.
Time Frame: Day 7
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Ibuprofen Capsule (400 mg) | Ibuprofen Tablet (400 mg) | Paracetamol Tablet (1000 mg) | Placebo Tablet
Number analyzed (Participants) | 23 | 22 | 27 | 23
Participants | 12 | 8 | 4 | 0
Statistical Analysis 1: Comparison: Ibuprofen Capsule (400 mg) vs Paracetamol Tablet (1000 mg); Test type: Superiority or Other; p = 0.0084, Chi-squared — P-value associated with chi-square testing odds ratio; Odds Ratio (OR) = 6.19, 95% CI 2-sided [1.60 to 23.97] — Odds Ratio from logistic regression model with treatment as factor and period as covariate
Statistical Analysis 2: Comparison: Ibuprofen Tablet (400 mg) vs Paracetamol Tablet (1000 mg); Test type: Superiority or Other; p = 0.0999, Chi-squared — P-value associated with chi-square testing odds ratio; Odds Ratio (OR) = 3.19, 95% CI 2-sided [0.80 to 12.74] — Odds Ratio from logistic regression model with treatment as factor and period as covariate
Statistical Analysis 3: Comparison: Ibuprofen Capsule (400 mg) vs Ibuprofen Tablet (400 mg); Test type: Superiority or Other; p = 0.2845, Chi-squared; Odds Ratio (OR) = 1.94, 95% CI 2-sided [0.58 to 6.50] — Odds Ratio from logistic regression model with treatment as factor and period as covariate

5. Secondary Outcome: Incidence of Fecal Occult Blood
Description: The incidence of fecal occult blood was recorded as a binary response (0 = no presence of blood; 1 = presence of blood).
Time Frame: Day 7
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- Ibuprofen Capsule (400 mg): Two ibuprofen capsules (400 mg/capsule), were administered TID, orally with water.
- Ibuprofen Tablet (400 mg): Two ibuprofen tablet (400 mg/tablet), were administered TID, orally with water.
Arm/Group | Paracetamol Tablet (1000 mg) | Ibuprofen Capsule (400 mg) | Ibuprofen Tablet (400 mg) | Placebo Tablet
Number analyzed (Participants) | 27 | 23 | 22 | 22
Participants
  Score 0 = no fecal occult blood | 27 | 23 | 22 | 22
  Score 1 = fecal occult blood present | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the investigational product, and until 5 days following last administration of the investigational product.
Arm/Group | Paracetamol Tablet (1000 mg) | Ibuprofen Capsule (400 mg) | Ibuprofen Tablet (400 mg) | Placebo Tablet
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/24 | 1/23 | 0/28
Other Adverse Events (participants affected / at risk) | 4/28 | 5/24 | 4/23 | 1/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paracetamol Tablet (1000 mg) (N=28) | Ibuprofen Capsule (400 mg) (N=24) | Ibuprofen Tablet (400 mg) (N=23) | Placebo Tablet (N=28)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paracetamol Tablet (1000 mg) (N=28) | Ibuprofen Capsule (400 mg) (N=24) | Ibuprofen Tablet (400 mg) (N=23) | Placebo Tablet (N=23)
Abdominal Pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.